CLINICAL TRIAL: NCT01579006
Title: A Multi National, Multi-center Non-interventional Study in Rheumatoid Arthritis (RA) Patients Treated With Tocilizumab (Actemra)
Brief Title: Observational Study of RoActemra/Actemra (Tocilizumab) in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Clalit Health Services (Other)
Responsible Party: Sponsor
Other Study IDs: ML28164
Record Dates: First submitted 2012-04-16; First posted 2012-04-17 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab
  Other Names: Actemra

SUMMARY:
This multi-center, observational study will evaluate the clinical practice patterns, efficacy and safety of RoActemra/Actemra in patients with rheumatoid arthritis who have had an inadequate response (or were intolerant to) treatment with non-biological DMARDs or with one biological agent. Data will be collected from each eligible patient initiated on RoActemra/Actemra treatment by their treating physician according to approved label for 6 months from start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Moderate to severe rheumatoid arthritis
* Inadequate response (or intolerant) to non-biological DMARDs or one biologic agent
* Patients initiating treatment with RoActemra/Actemra on their physician's decision (in accordance with the local label), including patients who started treatment with RoActemra/Actemra in the 8 weeks prior to the enrolment visit

Exclusion Criteria:

* RoActemra/Actemra treatment more than 8 weeks prior to the enrolment visit
* Previous RoActemra/Actemra treatment in a clinical trial or for compassionate use
* Enrolled in an ongoing clinical trial and/or treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational agent, whichever is longer) before starting treatment with RoActemra/Actemra
* History of autoimmune disease or any joint inflammatory disease other than rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients treated with tocilizumab
Sampling Method: Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2012-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- Israel (9):
  - Afula
  - Beer Yaakov
  - Beersheba
  - Hadera
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Ramat Gan

RESULTS

PARTICIPANT FLOW:
Groups:
- Rheumatoid Arthritis Participants: Participants with moderate to severe rheumatoid arthritis (RA), according to the American College of Rheumatology (ACR) criteria and the Disease Activity Score Based on 28 Joints (DAS28), who have had an inadequate response (or were intolerant) to treatment with non-biological disease-modifying anti-rheumatic drugs (DMARDs) or with one biological agent in whom the attending physician decided to start treatment with tocilizumab (TCZ) (according to local label) at the time of recruitment or up to 8 week prior to the time of recruitment were observed for 6 months.
Period: Overall Study
Arm/Group | Rheumatoid Arthritis Participants
Started | 184
Completed | 151
Not Completed | 33
Not completed — Lack of Efficacy | 10
Not completed — Adverse Event | 13
Not completed — Withdrawal by Subject | 5
Not completed — Non-compliance | 3
Not completed — Due to participant's health fund | 1
Not completed — Scheduled surgery | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) population included all recruited participants who received at least one dose of TCZ.
Groups:
- Rheumatoid Arthritis Participants: Participants with moderate to severe RA, according to the ACR criteria and the DAS28, who have had an inadequate response (or were intolerant) to treatment with non-biological DMARDs or with one biological agent in whom the attending physician decided to start treatment with TCZ (according to local label) at the time of recruitment or up to 8 week prior to the time of recruitment were observed for 6 months.
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141
  Male | 43

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants on TCZ Treatment at 6 Months After Treatment Initiation
Time Frame: 6 months
Population: FAS population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 184
percentage of participants | 42.4 [35.1542 to 49.8776]

2. Secondary Outcome: Percentage of Participants With Systemic Manifestations of RA at Baseline
Description: Systemic manifestations included fibromyalgia, osteoporosis, sjogren's syndrome, anemia, rheumatoid nodules, pulmonary fibrosis, vasculitis, peripheral neuropathy or mononeuropathy, scleritis, episcleritis, hypertension, hyperlipidemia, low high-density lipoproteins, diabetes type 1 and type 2, metabolic syndrome, carotid artery disease, transient ischemic attacks, embolic stroke, atherothrombotic stroke, atrial fibrillation, heart failure New York Heart Association (NYHA) Class l/ll, coronary heart disease(angina pectoris/myocardial), aortic aneurism, peripheral arterial occlusive disease, percutaneous coronary interventions, coronary artery bypass, carotid endarterectomy and peripheral arterial bypass.
Time Frame: Baseline
Population: FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 184
percentage of participants
  Fibromyalgia | 8.7
  Osteoporosis | 22.3
  Sjogren's syndrome | 6.5
  Anemia | 21.8
  Rheumatoid nodules | 8.1
  Pulmonary fibrosis | 3.2
  Vasculitis | 0.5
  Peripheral neuropathy or mononeuropathy | 4.3
  Scleritis | 1.6
  Episcleritis | 0.5
  Hypertension | 32.1
  Hyperlipidemia | 38.0
  Low high-density lipoproteins | 8.7
  Diabetes type 1 and type 2 | 15.2
  Metabolic syndrome | 10.3
  Carotid artery disease | 1.1
  Transient ischemic attacks | 3.3
  Embolic stroke | 0.5
  Atherothrombotic stroke | 2.7
  Atrial fibrillation | 1.1
  Heart Failure NYHA class l/ll | 1.6
  Coronary heart disease(angina pectoris/myocardial) | 6.0
  Aortic aneurism | 0.5
  Peripheral arterial occlusive disease | 0.5
  Percutaneous coronary interventions | 4.4
  Coronary artery bypass | 1.6
  Carotid Endarterectomy | 0.5
  Peripheral arterial bypass | 2.1

3. Secondary Outcome: Percentage of Participants Who Received DMARDs Prior to Start of Study and Concomitantly With TCZ During the Study
Description: DMARDs exposure was evaluated for all participants. "Prior DMARDs treatment" included participants, who were treated with DMARDs 8 weeks and according to physician's discretion before being included in the study. "DMARDs treatment at baseline" included participants who were receiving DMARDs when they were included in the study and continued with this concomitant medication in addition to TCZ. Only those participants who received DMARDs prior to start of study and at Baseline up to 6 months were reported.
Time Frame: Prior to study start (8 weeks) and Baseline up to 6 months
Population: FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 184
percentage of participants
  Azathioprine: Prior to study | 0.6
  Gold Compounds: Prior to study | 2.2
  Hydroxychloroquine: Prior to study | 33.3
  Leflunomide: Prior to study | 7.9
  Methotrexate: Prior to study | 24.5
  Sulfasalazine: Prior to study | 29.2
  Other DMARD: Prior to study | 2.2
  Azathioprine: Adm 1 to 6 | 1.1
  Gold Compounds: Adm 1 to 6 | 3.3
  Hydroxychloroquine: Adm 1 to 6 | 84.8
  Leflunomide: Adm 1 to 6 | 25.0
  Methotrexate: Adm 1 to 6 | 96.2
  Other DMARD: Adm 1 to 6 | 20.7
  Sulfasalazine: Adm 1 to 6 | 69.0

4. Secondary Outcome: Percentage of Participants With Reason for DMARD Withdrawal
Description: Objective intolerance was determined by medical observation; subjective intolerance was determined by the participant; lack of efficacy was determined by physician discretion.
Time Frame: Up to 6 months
Population: FAS population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 184
percentage of participants
  Methotrexate: Lack of efficacy | 27.3 [19.2170 to 36.5911]
  Methotrexate: Intolerance,Objective | 22.7 [15.2801 to 31.6955]
  Methotrexate: Intolerance,Subjective | 17.3 [10.7316 to 25.6520]
  Methotrexate: Other | 32.7 [24.0832 to 42.3279]
  Hydroxychloroquine: Lack of efficacy | 60.0 [50.4498 to 69.0222]
  Hydroxychloroquine: Intolerance,Objective | 14.8 [8.8536 to 22.6102]
  Hydroxychloroquine: Intolerance,Subjective | 12.2 [6.8181 to 19.5816]
  Hydroxychloroquine: Other | 13.0 [7.4878 to 20.5993]
  Sulfasalazine: Lack of efficacy | 60.6 [50.7331 to 69.7795]
  Sulfasalazine: Intolerance,Objective | 11.9 [6.5057 to 19.5311]
  Sulfasalazine: Intolerance,Subjective | 9.2 [4.4876 to 16.2252]
  Sulfasalazine: Other | 18.3 [11.5831 to 26.9055]
  Leflunomide: Lack of efficacy | 63.2 [45.9943 to 78.1875]
  Leflunomide: Intolerance,Objective | 5.3 [0.6439 to 17.7491]
  Leflunomide: Intolerance,Subjective | 10.5 [2.9435 to 24.8049]
  Leflunomide: Other | 21.1 [9.5541 to 37.3188]
  Gold compounds: Lack of efficacy | 100 [66.3733 to 100.0000]
  Azathioprine: Lack of efficacy | 66.7 [9.4299 to 99.1596]
  Azathioprine: Intolerance, Subjective | 33.3 [0.8404 to 90.5701]
  Other: Lack of efficacy | 44.0 [24.4024 to 65.0718]
  Other: Intolerance,Objective | 8.0 [0.9840 to 26.0306]
  Other: Intolerance,Subjective | 16.0 [4.5379 to 36.0828]
  Other: Unspecified | 32.0 [14.9495 to 53.5001]

5. Secondary Outcome: Percentage of Participants Who Received Biological RA Treatment Prior to Start of Study
Description: Biological RA treatment exposure was evaluated for all participants. "Prior biological RA treatment" included participants who were treated with biological RA treatment 8 weeks before being included in the study. Percentage of participants who did not receive any biological RA treatment and percentage of participants who received one or more biologic RA treatments were reported.
Time Frame: Prior to study start (8 weeks)
Population: FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 184
percentage of participants
  Did not receive any biologic RA treatment | 53.8
  Received 1 biologic RA treatment | 38.6
  Received 2 biologic RA treatments | 7.1
  Received 3 or more biologic RA treatments | 0.5

6. Secondary Outcome: Percentage of Participants With Type of Previous Biologic RA Treatments
Description: Previous biologic RA treatment included adalimumab, infliximab, golimumab, etanercept, certolizumab, and other (any other previous biologic RA treatment). Same participants may be counted in more than one previous biologic RA treatment category.
Time Frame: Up to 6 months
Population: FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 184
percentage of participants
  Adalimumab | 15.2
  Infliximab | 8.2
  Golimumab | 4.3
  Etanercept | 17.4
  Certolizumab | 1.6
  Other | 7.6

7. Secondary Outcome: Duration of Previous Biologic RA Treatments
Description: Previous biologic RA treatment included adalimumab, infliximab, golimumab, etanercept, certolizumab, and other (any other previous biologic RA treatment).
Time Frame: Up to 6 months
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure and "n"= participants who were evaluable for each category.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 85
years
  Adalimumab (n=27) | 0.9 (1.0)
  Infliximab (n=14) | 2.5 (2.9)
  Golimumab (n=8) | 1.6 (0.8)
  Etanercept (n=31) | 1.7 (1.9)
  Certolizumab (n=3) | 4.9 (1.9)
  Other (n=13) | 1.4 (2.2)

8. Secondary Outcome: Percentage of Participants With Reasons for Termination of Previous Biologic RA Treatments
Description: Lack of efficacy was determined by physician discretion. Previous biologic RA treatment included adalimumab, infliximab, golimumab, etanercept, certolizumab, and other (any other previous biologic RA treatment).
Time Frame: Up to 6 months
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 184
percentage of participants
  Adalimumab: Lack of efficacy (n=28) | 85.7
  Adalimumab: Adverse event (n=28) | 10.7
  Adalimumab: Other (n=28) | 3.6
  Infliximab: Lack of efficacy (n=15) | 53.3
  Infliximab: Adverse event (n=15) | 26.7
  Infliximab: Other (n=15) | 20.0
  Golimumab: Lack of efficacy (n=8) | 62.5
  Golimumab: Adverse event (n=8) | 25.0
  Golimumab: Other (n=8) | 12.5
  Etanercept: Lack of efficacy (n=31) | 67.7
  Etanercept: Adverse event (n=31) | 19.4
  Etanercept: Other (n=31) | 12.9
  Certolizumab: Lack of efficacy (n=3) | 33.3
  Certolizumab: Adverse event (n=3) | 33.3
  Certolizumab: Other (n=3) | 33.3
  Other: Lack of efficacy (n=13) | 53.8
  Other: Adverse event (n=13) | 15.4
  Other: Unspecified (n=13) | 30.8

9. Secondary Outcome: Percentage of Participants With Dose Modifications
Description: TCZ was administered every 4 weeks according to the label. Due to the observational nature of the study, the suggested schedule was subject to changes according to physician and participant considerations.
Time Frame: 6 months
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 183
percentage of participants
  TCZ Administration 1 (Baseline) (n=183) | 0.0 [0.0000 to 1.9956]
  TCZ Administration 2 (Week 4) (n=178) | 2.8 [0.9182 to 6.4332]
  TCZ Administration 3 (Week 8) (n=174) | 2.3 [0.6298 to 5.7811]
  TCZ Administration 4 (Week 12) (n=166) | 1.8 [0.3743 to 5.1904]
  TCZ Administration 5 (Week 16) (n=158) | 1.9 [0.3933 to 5.4484]
  TCZ Administration 6 (Week 20) (n=151) | 3.3 [1.0837 to 7.5580]

10. Secondary Outcome: Percentage of Participants With Reasons for Dose Modification
Description: TCZ was administered every 4 weeks according to the label. Due to the observational nature of the study, the suggested schedule was subject to changes according to physician and participant considerations. Only those participants who had dose modifications were reported.
Time Frame: 6 months
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 20
percentage of participants
  TCZ Administration 2 (Week 4):Adverse event/safety | 80.0 [28.3582 to 99.4949]
  TCZ Administration 2 (Week 4):Other reason | 20.0 [0.5051 to 71.6418]
  TCZ Administration 3 (Week 8):Adverse event/safety | 100.0 [39.7635 to 100.0000]
  TCZ Administration 4(Week 12):Adverse event/safety | 66.7 [9.4299 to 99.1596]
  TCZ Administration 4 (Week 12): Other reason | 33.3 [0.8404 to 90.5701]
  TCZ Administration 5(Week 16):Adverse event/safety | 100.0 [29.2402 to 100.0000]
  TCZ Administration 6(Week 20):Adverse event/safety | 40.0 [5.2745 to 85.3367]
  TCZ Administration 6 (Week 20): Other reason | 60.0 [14.6633 to 94.7255]

11. Secondary Outcome: Mean Dose at 6 Months
Description: as for outcome 9
Time Frame: 6 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milligrams per kilogram (mg/kg)
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 182
milligrams per kilogram (mg/kg)
  TCZ Administration 1 (Baseline) (n=182) | 8.0 (0.0)
  TCZ Administration 2 (Week 4) (n=179) | 7.9 (0.6)
  TCZ Administration 3 (Week 8) (n=174) | 7.9 (0.6)
  TCZ Administration 4 (Week 12) (n=166) | 7.9 (0.5)
  TCZ Administration 5 (Week 16) (n=158) | 7.9 (0.3)
  TCZ Administration 6 (Week 20) (n=151) | 7.9 (0.5)

12. Secondary Outcome: Mean Number of Dose Modifications at 6 Months
Description: as for outcome 9
Time Frame: 6 months
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: dose modification
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 12
dose modification | 1.7 (0.9)

13. Secondary Outcome: Mean Dosing Interval of Treatment at 6 Months
Description: TCZ was administered every 4 weeks according to the label. Due to the observational nature of the study, the suggested schedule was subject to changes according to physician and participant considerations. The mean dosing interval between different TCZ administrations (Adm) by participants within 6 months observational period was presented.
Time Frame: 6 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 178
days
  Between TCZ Adm 1 (Baseline) and 2 (Week 4)(n=178) | 31.4 (5.7)
  Between TCZ Adm 2 (Week 4) and 3 (Week 8) (n=174) | 30.8 (4.5)
  Between TCZ Adm 3 (Week 8) and 4 (Week 12) (n=166) | 31.4 (4.7)
  Between TCZ Adm 4 (Week 12) and 5 (Week 16)(n=158) | 31.8 (7.2)
  Between TCZ Adm 5 (Week 16) and 6 (Week 20)(n=150) | 31.9 (8.6)

14. Secondary Outcome: Percentage of Participants Who Discontinued From TCZ for Safety Versus Efficacy
Description: The safety variable measured the number of participants who discontinued TCZ due to adverse reactions to TCZ, and the efficacy variable measured the participants who discontinued from TCZ due to lack of efficacy according to criteria of the treating physician.
Time Frame: 6 months
Population: FAS population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 184
percentage of participants
  Lack of efficacy | 6.0 [3.0218 to 10.4448]
  Adverse event | 6.5 [3.4150 to 11.1150]
  Other | 5.4 [2.6366 to 9.7675]

15. Secondary Outcome: Time to Restoration of Initial Dosing Regimen
Time Frame: 6 months
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 7
days | 81.6 (34.9)

16. Secondary Outcome: Percentage of Participants Who Adhered to the Dosing Regimen Recommended by Physician
Description: A participant's adherence was calculated based on the adverse event or laboratory abnormality experienced by the participants who required dose modifications as per local TCZ label or protocol.
Time Frame: 6 months
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 15
percentage of participants | 8.2 [4.6345 to 13.0893]

17. Secondary Outcome: Percentage of Participants on TCZ Monotherapy
Description: TCZ was administered every 4 weeks according to the label. Due to the observational nature of the study, the suggested schedule was subject to changes according to physician and participant considerations. Only those participants who had TCZ as monotherapy were reported.
Time Frame: Up to 6 months
Population: FAS population. Here, "n"= participants who were evaluable for each category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 184
percentage of participants
  TCZ Administration 1 (Baseline) (n=184) | 32.6 [25.8944 to 39.8940]
  TCZ Administration 2 (Week 4) (n=178) | 34.3 [27.3324 to 41.7408]
  TCZ Administration 3 (Week 8) (n=174) | 35.6 [28.5300 to 43.2332]
  TCZ Administration 4 (Week 12) (n=166) | 38.0 [30.5448 to 45.7972]
  TCZ Administration 5 (Week 16) (n=158) | 38.6 [30.9797 to 46.6713]
  TCZ Administration 6 (Week 20) (n=151) | 41.7 [33.7596 to 50.0155]

18. Secondary Outcome: Change From Baseline in Tender Joint Count (TJC) (68 Joints) at Month 6
Description: The number of tender joints was recorded on the joint assessment form, with no tenderness = 0, and tenderness = 1, for 68 joints, giving a total possible TJC score of 0 to 68.
Time Frame: Baseline, 6 months
Population: FAS population. Here, number of participants analyzed = participants with valid data to calculate TJC at the end of study (6 months).
Measure: Mean (Standard Deviation); unit: Tender Joint Count
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 67
Tender Joint Count | -10.7 (10.3)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank Test

19. Secondary Outcome: Change From Baseline in Swollen Joint Count (SJC) (66 Joints) at Month 6
Description: The number of swollen joints was recorded on the joint assessment form, with no swelling = 0, and swelling =1, for 66 joints, giving a total possible SJC score of 0 to 66.
Time Frame: Baseline, 6 months
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Swollen Joint Count
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 67
Swollen Joint Count | -6.7 (7.5)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank Test

20. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28 Joints (DAS28) at Month 6
Description: DAS28 was calculated from SJC and TJC using an assessment of 28 joints, the erythrocyte sedimentation rate (ESR) (milliliter per hour [mm/hr]), and Patient's Global Assessment (PGH) of disease activity (measured on a 0 to 100 mm Visual Analogue Scale [VAS] where 0=no disease activity and 100=worst disease activity). DAS28 was calculated using the following formula: DAS28 = 0.56*square root (sqrt) (TJC28) + 0.28*sqrt(SJC28) + 0.70*natural logarithm (ln) (ESR) + 0.014*PGH of disease activity. Total score range: 0-10, with a higher score indicated more disease activity. DAS28 <=3.2 implied low disease activity, DAS >3.2 to 5.1 implied moderate disease activity and DAS >5.1 implied high disease activity, and DAS28 <2.6 = clinical remission.
Time Frame: Baseline, 6 months
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 46
Score on a scale | -2.7 (1.7)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank Test

21. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR) Response at Month 6
Description: Clinical response assessed as per EULAR categorical DAS28 response criteria was defined as clinically meaningful improvement at a particular time point. EULAR response was based on change from baseline (CFB) in the DAS28 score and also on the actual DAS28 score at the time point so was more reflective of the current status of the participant. The DAS28 score was a measure of the participant's disease activity, based on the TJC (28 joints), SJC (28 joints), PGH (mm), and ESR (mm/hr). DAS28 total scores ranged from 0 to approximately 10. Scores <2.6 = best disease control and scores >5.1 = worse disease control. A negative CFB indicated clinically meaningful improvement. EULAR Good response: DAS28 <=3.2 and a CFB <-1.2. EULAR Moderate response: DAS28 >3.2 to ≤ 5.1 or a CFB < -0.6 to ≥ -1.2. EULAR No response: DAS28 ≤3.2 or CFB >=-0.6, DAS28 >3.2 to <=5.1 or CFB >=-0.6 and DAS28 >5.1 or CFB >=-0.6.
Time Frame: 6 months
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 46
percentage of participants
  Good | 56.5 [41.1071 to 71.0657]
  Moderate | 28.3 [15.9867 to 43.4604]
  No response | 15.2 [6.3444 to 28.8691]

22. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) Score at Month 6
Description: The SDAI was a combined index for measuring disease activity in RA which reflected the numerical sum of five outcome parameters: TJC and SJC based on a 28-joint assessment, PGH and physician's global assessment (PhGH) of disease activity, assessed on 0-100 mm VAS where 0 = no disease activity and 100 = worst disease activity, and C-reactive protein (CRP) (milligrams per deciliter [mg/dL]). SDAI total score = 0-86. A SDAI score of <=3.3 represented clinical remission, a score of <=11.0 represents low disease activity, a score of <=26.0 represented moderate disease activity and a score of >26.0 represented high (or severe) disease.
Time Frame: Baseline, 6 months
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 52
Score on a scale | -18.7 (16.7)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank Test

23. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) Score at Month 6
Description: The CDAI was a combined index for measuring disease activity in RA and used to evaluate disease activity in the absence of laboratory testing of CRP and ESR. It was the numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, PGH and PhGH (assessed on 0-100 mm); VAS (0 = no disease activity and 100 = worst disease activity). CDAI total score = 0-76. A CDAI score of <=2.8 represented clinical remission, a score of <=10.0 represented low disease activity, a score of <=22.0 represented moderate disease activity and a score of >22.0 represented high (or severe) disease.
Time Frame: Baseline, 6 months
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 70
Score on a scale | -17.3 (15.2)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank Test

24. Secondary Outcome: Percentage of Participants Who Achieved 20% Improvement in ACR (ACR20) Response at Month 6
Description: ACR response was calculated based on total joint count evaluation (28 or 66/68 joint count) and other clinical and laboratory assessments. A positive ACR20 response required at least a 20% improvement (reduction) compared to baseline in swollen joint count (66 joints) and tender joint count (68 joints) and at least 3 of the following 5 assessments: participant's global assessment of pain, PGH, PhGH (all 3 assessed at 0 [good] to 100 mm [worst] VAS scale), participant assessment of disability measured by the Health Assessment Questionnaire-Disability Index (HAQ-DI) (assessed on a 0 to 3 scale, where higher scores represented higher disease activity), Acute phase reactant (CRP or ESR). A reduction in the level of and acute phase reactants was considered an improvement.
Time Frame: 6 months
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 31
percentage of participants | 54.8

25. Secondary Outcome: Percentage of Participants Who Achieved 50% Improvement in ACR (ACR50) Response at Month 6
Description: ACR response was calculated based on total joint count evaluation (28 or 66/68 joint count) and other clinical and laboratory assessments. A positive ACR50 response required at least a 50% improvement (reduction) compared to baseline in swollen joint count (66 joints) and tender joint count (68 joints) and at least 3 of the following 5 assessments: (participant's global assessment of pain, PGH, PhGH (all 3 assessed at 0 [good] to 100 mm [worst] VAS scale), participant assessment of disability measured by the Health Assessment Questionnaire-Disability Index (HAQ-DI) (assessed on a 0 to 3 scale, where higher scores represented higher disease activity), and acute phase reactant (CRP or ESR). A reduction in the level of acute phase reactants was considered an improvement.
Time Frame: 6 months
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 31
percentage of participants | 32.3

26. Secondary Outcome: Percentage of Participants Who Achieved 70% Improvement in ACR (ACR70) Response at Month 6
Description: ACR response was calculated based on total joint count evaluation (28 or 66/68 joint count) and other clinical and laboratory assessments. A positive ACR70 response required at least a 70% improvement (reduction) compared to baseline in swollen joint count (66 joints) and tender joint count (68 joints) and at least 3 of the following 5 assessments: (participant's global assessment of pain, PGH, PhGH (all 3 assessed at 0 [good] to 100 mm [worst] VAS scale), participant assessment of disability measured by the Health Assessment Questionnaire-Disability Index (HAQ-DI) (assessed on a 0 to 3 scale, where higher scores represented higher disease activity), and acute phase reactant (CRP or ESR). A reduction in the level of acute phase reactants was considered an improvement.
Time Frame: 6 months
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 31
percentage of participants | 9.7

27. Secondary Outcome: Change From Baseline in CRP at Month 6
Description: The test for CRP was a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. The serum concentration of CRP was measured in mg/dL. A reduction in the level was considered an improvement.
Time Frame: Baseline, 6 months
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 55
mg/dL | -1.6 (2.5)

28. Secondary Outcome: Change From Baseline in ESR at Month 6
Description: ESR was a laboratory test that provided a non-specific measure of inflammation. The test assessed the rate at which red blood cells fell in a test tube. ESR was measured in mm/hr. A reduction in the level was considered an improvement.
Time Frame: Baseline, 6 months
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 49
mm/hr | -34.4 (26.1)

29. Secondary Outcome: Change From Baseline in PhGH at Month 6
Description: The PhGH was assessed using a 0 to 100 mm horizontal VAS by the physician. The left-hand extreme of the line equaled 0 mm, and was described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equaled 100 mm, as "maximum disease activity" (maximum arthritis disease activity). A negative change from baseline indicated improvement.
Time Frame: Baseline, 6 months
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 72
mm | -34.0 (28.2)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank Test

30. Secondary Outcome: Change From Baseline in PGH of Disease Activity at Month 6
Description: The PGH of disease activity was assessed using a 0 to 100 mm horizontal VAS by the participant. The left-hand extreme of the line equaled 0 mm, and was described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equaled 100 mm, as "maximum disease activity" (maximum arthritis disease activity). A negative change from baseline indicated improvement.
Time Frame: Baseline, 6 months
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 75
mm | -26.5 (28.4)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank Test

31. Secondary Outcome: Change From Baseline in HAQ-DI at Month 6
Description: The HAQ-DI was a participant self-reported questionnaire for assessing the extent of a participant's functional ability. It consisted of 20 questions in 8 categories (dressing and grooming, rising, eating, walking, reach, grip, hygiene, and carrying out daily activities). Each question had 4 response options, ranging from "no difficulty" to "unable to do", corresponding to scores from 0 to 3. The HAQ-DI scale was an average of all the scores and ranged from 0 to 3, where higher scores represented higher disease activity. A score of <0.5 represented clinical remission. A participant achieved a clinically meaningful improvement in HAQ-DI if they had a reduction from baseline of >=0.22.
Time Frame: Baseline, 6 months
Population: ITT population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 77
Score on a scale | -0.3 (0.7)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank Test

32. Secondary Outcome: Change From Baseline in Participant's Assessment of Fatigue Using VAS at Month 6
Description: Fatigue was evaluated by a VAS. Participants marked on a 100 mm horizontal VAS the level of fatigue that they have experienced, ranging from 0 (no fatigue) to 100 (extreme fatigue).
Time Frame: Baseline, 6 months
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 74
mm | -17.9 (31.1)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank Test

33. Secondary Outcome: Change From Baseline in Participant's Assessment of RA-Related Pain at Month 6
Description: Severity of pain was evaluated by a VAS. Participants marked on a 100 mm horizontal VAS the severity of pain that they had experienced because of their RA, ranging from 0 (no pain) to 100 (unbearable pain). A decrease of 10 points was considered clinically meaningful.
Time Frame: Baseline, 6 months
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 76
mm | -23.7 (32.6)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank Test

34. Secondary Outcome: Change From Administration 1 in Functional Assessment of Chronic Illness Therapy (FACIT)- Fatigue Questionnaire at Month 6
Description: The FACIT Measurement System was a collection of health-related quality of life questionnaires targeted to the management of chronic illness and included questions on Physical Well-Being, Social/Family Well-Being, Emotional Well-Being and Functional Well-Being. The FACIT Fatigue Scale was a 13-item tool that measured an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue was measured on a five-point Likert scale (4 = not at all fatigued to 0 = very much fatigued). The total score of FACIT ranged from 0 to 160. An increase of 4 points in the FACIT-Fatigue score was considered clinically meaningful. Change from Administration 1 was reported for individual administration schedules. TCZ was administered every 4 weeks according to the label. Due to the observational nature of the study, the suggested schedule was subject to changes according to physician and participant considerations.
Time Frame: Administration 1 (Baseline), 6 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 55
Score on a scale
  Change at Administration 2 (n=38) | 7.3 (12.7)
  Change at Administration 3 (n=39) | 11.7 (18.1)
  Change at Administration 4 (n=35) | 11.9 (18.3)
  Change at Administration 5 (n=31) | 17.3 (20.5)
  Change at Administration 6 (n=33) | 20.0 (23.9)

35. Secondary Outcome: Change From Baseline in Morning Stiffness as Assessed Using VAS at Month 6
Description: Morning stiffness was defined by the time elapsed between the time of usual awakening (even if not in the morning) and the time the participant was as limber as he/she would be during a day involving typical activities. Morning stiffness was assessed on a 100 mm VAS, where 0= none and 100= very severe.
Time Frame: Baseline, 6 months
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 76
mm | -26.6 (34.9)
Statistical Analysis 1: Comparison: Rheumatoid Arthritis Participants; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank Test

36. Primary Outcome: Percentage of Participants on TCZ Treatment at 5-6 Months After Treatment Initiation
Time Frame: 5-6 months
Population: FAS population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 184
percentage of participants | 85.9 [79.9850 to 90.5573]

ADVERSE EVENTS:
Time Frame: Up to 6 months
Groups:
- Rheumatoid Arthritis Participants: Participants with moderate to severe RA, according to the ACR criteria and the DAS28, who had been receiving TCZ in the past and in whom the attending physician decided to start treatment with TCZ at the time of recruitment (according to the local label) were observed for 6 months.
Arm/Group | Rheumatoid Arthritis Participants
Serious Adverse Events (participants affected / at risk) | 17/184
Other Adverse Events (participants affected / at risk) | 77/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rheumatoid Arthritis Participants (N=184)
Microcytic anaemia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Upper abdominal pain (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Pneumonia (Infections and infestations) | 1
Post procedural sepsis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Acute renal failure (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rheumatoid Arthritis Participants (N=184)
Anaemia (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 5
Lymphocytosis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 3
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Oral pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Malaise (General disorders) | 1
Pyrexia (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Gingival infection (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Arteriogram coronary (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood thyroid stimulating hormone increased (Investigations) | 1
Blood triglycerides increased (Investigations) | 1
Full blood count decreased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 6
Liver function test abnormal (Investigations) | 2
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Transaminases increased (Investigations) | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 2
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2
Hirsutism (Skin and subcutaneous tissue disorders) | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.